CLINICAL TRIAL: NCT06946251
Title: Evaluation of Patients With Reduced and Preserved Ejection Fraction After Transcutaneous Diaphragm Stimulation
Brief Title: Transcutaneous Diaphragm Stimulation in ICU Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, A. Oguzhan KUCUK, MD, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/9
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Patients
Keywords: Diaphragm Stimulation; Intensive care unit; Ejection Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Patients with low EF who receive TEDS (Experimental)
  Interventions: Device: Transcutaneous Diaphragm Stimulation
- Group 2: Patients with high EF who receive TEDS (Experimental)
  Interventions: Device: Transcutaneous Diaphragm Stimulation
- Group 3: Patients with low EF who do not receive TEDS (No Intervention)
- Group 4: Patients with high EF who do not receive TEDS (No Intervention)

INTERVENTIONS:
Device: Transcutaneous Diaphragm Stimulation — In the ICU, TEDS is administered by a physiotherapist once daily for 20 minutes, five days a week, as part of the routine treatment protocol. The stimulation is delivered using the LGT-231 model device from the LONGEST brand.
  A transcutaneous current with a frequency of 30-50 Hz and a pulse width of 300-400 microseconds is applied to the diaphragm. The stimulation intensity is increased until visible muscle contraction is achieved.
  Arms: Group 1: Patients with low EF who receive TEDS; Group 2: Patients with high EF who receive TEDS

SUMMARY:
The aim of this study is to compare the effects of transcutaneous electrical diaphragm stimulation (TEDS) on diaphragm thickness, duration of mechanical ventilation, length of ICU stay, and right/left heart functions between patient groups with low and high ejection fraction (EF) levels.

This randomized controlled trial will record demographic data, diaphragm ultrasound measurements, and echocardiographic findings of patients who receive or do not receive TEDS for five consecutive days.

Participants will be divided into four groups according to their EF levels and whether or not they receive diaphragm stimulation:

Group 1: Patients with low EF who receive TEDS Group 2: Patients with high EF who receive TEDS Group 3: Patients with low EF who do not receive TEDS Group 4: Patients with high EF who do not receive TEDS

Diaphragm thickness and echocardiographic assessments will be performed at baseline and at the end of the five-day TEDS intervention.

TEDS Application Protocol

In the ICU, TEDS is administered by a physiotherapist once daily for 20 minutes, five days a week, as part of the routine treatment protocol. The stimulation is delivered using the LGT-231 model device from the LONGEST brand.

A transcutaneous current with a frequency of 30-50 Hz and a pulse width of 300-400 microseconds is applied to the diaphragm. The stimulation intensity is increased until visible muscle contraction is achieved.

Electrode placement involves:

The first pair of electrodes placed bilaterally between the 8th and 10th anterior intercostal spaces, lateral to the xiphoid process.

The second pair placed along the mid-axillary line of the thorax, also between the 8th and 10th intercostal spaces.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years
* Patients expected to require mechanical ventilation for at least 72 hours

Exclusion Criteria:

* Presence of known neuromuscular diseases that contraindicate the use of transcutaneous diaphragm stimulation
* Phrenic nerve injury
* History of abdominal or thoracic surgery that prevents the application of diaphragm stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Diaphragm Thickness and Thickening Fraction Measured by Ultrasound | At baseline (Day 0) and on Day 5 of the study
  Diaphragm thickness will be measured using B-mode ultrasonography. The following parameters will be assessed:
  Diaphragm thickness at end-expiration (Tdi-exp), in millimeters (mm)
  Diaphragm thickness at end-inspiration (Tdi-insp), in millimeters (mm)
  Diaphragm thickening fraction (TF), calculated using the following formula:
  TF = (Tdi-insp - Tdi-exp) / Tdi-exp × 100.
Duration of mechanical ventilation | At the beginning of the study and at the end of the 5-day period
  Length of ICU stay will be recorded in days for each patient during the 5-day study follow-up. The duration will be calculated from the date and time of ICU admission until discharge or the end of the 5-day observation period, whichever comes first. Data will be obtained from patient medical records.
Length of stay in the intensive care unit | At the beginning of the study and at the end of the 5-day period
  The total number of days each patient remains in the intensive care unit (ICU) will be recorded during the 5-day follow-up period. ICU stay duration will be calculated from the time of ICU admission until ICU discharge or the end of the 5-day observation period, whichever occurs first. Data will be obtained from patient medical records.
Cardiac Function Parameters Assessed by Transthoracic Echocardiography | At baseline (Day 0) and on Day 5 of the study
  Cardiac function will be assessed using transthoracic echocardiography (TTE) performed by an experienced cardiologist. The following echocardiographic parameters will be recorded to evaluate both systolic and diastolic cardiac function:
  E/A ratio (m/s) e' velocity (cm/s) E/e' ratio Pulmonary vein flow pattern Peak flow velocity (m/s) Left atrial volume index (mL/m²) Left ventricular ejection fraction (LVEF, %) Right atrial volume (mL) Right ventricular volume (mL) Pulse Doppler myocardial performance index (RIMP) Tissue Doppler myocardial performance index (RIMP) Fractional area change (FAC, %) Tricuspid annular plane systolic excursion (TAPSE, cm) Tissue Doppler S wave velocity (cm/s)